CLINICAL TRIAL: NCT00623441
Title: E-Five Registry: To Evaluate the 'Real World' Clinical Performance of the Medtronic Endeavor ABT-578 Eluting Coronary Stent System; A Prospective, Multicenter Registry
Brief Title: E-Five Registry: A World-Wide Registry With The Endeavor Zotarolimus Eluting Coronary Stent
Acronym: eFive
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: Protocol Final version1.1; NCT00265668 (obsolete NCT alias)
Record Dates: First submitted 2008-02-18; First posted 2008-02-26 (Estimated); Results first posted 2011-12-16 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Endeavor Zotarolimus Eluting Coronary Stent — Drug eluting stent
  Other Names: Endeavor Stent

SUMMARY:
The safety and efficacy of the Endeavor(TM) ABT-578 Eluting Coronary Stent System has been assessed in a series of studies. The stent is coated with a proprietary drug compound that is designed to reduce restenosis.

This prospective multi-center study has been initiated:

* To document the acute and mid-term safety and overall clinical performance of the stent system in a "real world" patient population requiring stent implantation.
* To assess the event rate in patient subgroups with specific clinical indications and/or vessel or lesion characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >18 years of age (or minimum age as required by local regulation)
* The patient has consented to participate by signing the "Patient Informed Consent Form" and/or has authorized the collection and release of his medical information by signing the "Patient Data Release Consent Form".
* The patient is suitable for implantation of one or more Endeavor(TM) ABT-578 Eluting Coronary Stent System in one or more native artery target lesions.
* Lesion length and vessel diameter of the target lesion(s) are according to the "Indications for Use" as mentioned in the "Instructions for Use" that comes with every Endeavor(TM) ABT-578 Eluting Coronary Stent System.
* The patient is willing and able to cooperate with registry procedures and required follow up visits.

Exclusion Criteria:

* Women with known pregnancy or who are lactating.
* Patients with hypersensitivity or allergies to aspirin, heparin, clopidogrel, ticlopidine, drugs such as ABT-578, rapamycin, tacrolimus, sirolimus or similar drugs, or any other analogue or derivative, cobalt, chromium, nickel, molybdenum or contrast media.
* Patients in whom anti-platelet and/pr anticoagulation therapy is contraindicated.
* Patients who are judged to have a lesion that prevents complete inflation of an angioplasty balloon.
* Current medical condition with a life expectancy of less than 12 months.
* The subject is participating in another device or drug study. Subject must have completed the follow-up phase of any previous study at least 30 days prior to enrollment in this trial. The subject may only be enrolled in this E-five registry once.
* Patients with medical conditions that preclude the follow-up as defined in the protocol or that otherwise limits participation in this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-world patients requiring drug eluting stent implantation
Sampling Method: Non-Probability Sample
Enrollment: 8314 (Actual)
Dates: Start 2005-09; Primary Completion 2007-11 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian T Meredith, MD, Principal Investigator — Monash Medical Centre, Melbourne, Australia; Chaim Lotan, MD, Principal Investigator — Hadassah University Hospital, Jerusalem, Israel; Martin T Rothman, MD, Principal Investigator — London Chest Hospital, London, United Kingdom

REFERENCES:
- [Background] Fajadet J, Wijns W, Laarman GJ, Kuck KH, Ormiston J, Munzel T, Popma JJ, Fitzgerald PJ, Bonan R, Kuntz RE; ENDEAVOR II Investigators. Randomized, double-blind, multicenter study of the Endeavor zotarolimus-eluting phosphorylcholine-encapsulated stent for treatment of native coronary artery lesions: clinical and angiographic results of the ENDEAVOR II trial. Circulation. 2006 Aug 22;114(8):798-806. doi: 10.1161/CIRCULATIONAHA.105.591206. Epub 2006 Aug 14. PMID 16908773
- [Result] Jain AK, Meredith IT, Lotan C, Rothman MT, Pateraki S; E-Five Investigators. Real-world safety and efficacy of the endeavor zotarolimus-eluting stent: early data from the E-Five Registry. Am J Cardiol. 2007 Oct 22;100(8B):77M-83M. doi: 10.1016/j.amjcard.2007.08.026. PMID 17950836
- [Result] Lotan C, Meredith IT, Mauri L, Liu M, Rothman MT; E-Five Investigators. Safety and effectiveness of the Endeavor zotarolimus-eluting stent in real-world clinical practice: 12-month data from the E-Five registry. JACC Cardiovasc Interv. 2009 Dec;2(12):1227-35. doi: 10.1016/j.jcin.2009.10.001. PMID 20129549
- [Result] Jain AK, Lotan C, Meredith IT, Feres F, Zambahari R, Sinha N, Rothman MT; E-Five Registry Investigators. Twelve-month outcomes in patients with diabetes implanted with a zotarolimus-eluting stent: results from the E-Five Registry. Heart. 2010 Jun;96(11):848-53. doi: 10.1136/hrt.2009.184150. PMID 20478863
- [Result] Meredith I, Rothman M, Erglis A, Parikh K, Lotan C; E-Five Investigators. Extended follow-up safety and effectiveness of the Endeavor zotarolimus-eluting stent in real-world clinical practice: two-year follow-up from the E-Five Registry. Catheter Cardiovasc Interv. 2011 Jun 1;77(7):993-1000. doi: 10.1002/ccd.22803. Epub 2010 Dec 3. PMID 20853351
- [Result] Lotan C, Meredith IT, Jain A, Feres F, Firszt A, Garcia AF, Rothman MT. Clinical outcomes by geographic region for patients implanted with the zotarolimus-eluting stent. Arq Bras Cardiol. 2011 May;96(5):353-62. doi: 10.1590/s0066-782x2011005000033. Epub 2011 Apr 1. English, Portuguese, Spanish. PMID 21468534
- [Derived] Remak E, Manson S, Hutton J, Brasseur P, Olivier E, Gershlick A. Cost-effectiveness of the Endeavor stent in de novo native coronary artery lesions updated with contemporary data. EuroIntervention. 2010 Feb;5(7):826-32. doi: 10.4244/eijv5i7a138. PMID 20142198
- [Derived] Kandzari DE, Leon MB, Popma JJ, Fitzgerald PJ, O'Shaughnessy C, Ball MW, Turco M, Applegate RJ, Gurbel PA, Midei MG, Badre SS, Mauri L, Thompson KP, LeNarz LA, Kuntz RE; ENDEAVOR III Investigators. Comparison of zotarolimus-eluting and sirolimus-eluting stents in patients with native coronary artery disease: a randomized controlled trial. J Am Coll Cardiol. 2006 Dec 19;48(12):2440-7. doi: 10.1016/j.jacc.2006.08.035. Epub 2006 Nov 28. PMID 17174180
- See also: Related Info — http://www.medtronic.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive patients with an indication for coronary stent implantation according to the Instructions For Use of the Endeavor Coronary Stent, in whom it is an intent to implant one or more Endeavor Coronary Stents should be included (provided patient consent).
Pre-assignment Details: All enrolled subjects were followed for 12 months. An extended 2-year follow-up was performed in 2116 subjects from 26 centers.
Groups:
- Endeavor Coronary Stent: Patients with an indication for a percutaneous coronary intervention with implantation with a drug eluting stent
Period: Overall Study
Arm/Group | Endeavor Coronary Stent
Started | 8314
Completed | 8314 (12 months follow-up compliance was 94.2%)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Endeavor Coronary Stent
Number analyzed (Participants) | 8314
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4266
  >=65 years | 4048
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.29 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1940
  Male | 6374
Region of Enrollment [Number; unit: participants]
  Europe | 6566
  Southeast Asia | 879
  Pacifica | 57
  South America | 220
  Africa | 6
  India | 586
Diabetes Mellitus [Number; unit: Participants]
  IDDM (Insulin Dependent Diabetes Mellitus) | 682
  Non-IDDM (Non-Insulin Dependent Diabetes Mellitus) | 2039
  No Diabetes Mellitus | 5593

OUTCOME MEASURES:

1. Primary Outcome: MACE (Major Adverse Cardiac Events)
Description: MACE is defined as death, myocardial infarction (Q-wave and non-Q wave), emergent cardiac bypass surgery, or target lesion revascularization (repeat PTCA (Percutaneous Transluminal Coronary Angioplasty) or CABG (Coronary Artery Bypass Graft surgery))
Time Frame: 12 Months
Population: Intention to Treat (ITT)
Measure: Number; unit: Percentage of participants
Arm/Group | Endeavor Coronary Stent
Number analyzed (Participants) | 8314
Percentage of participants | 7.5

ADVERSE EVENTS:
Arm/Group | Endeavor Coronary Stent
Serious Adverse Events (participants affected / at risk) | 135/7832
Other Adverse Events (participants affected / at risk) | 0/7832
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endeavor Coronary Stent (N=7832)
Cardiac Death (Cardiac disorders) | 135 (135)

LIMITATIONS AND CAVEATS:
Data collection in this large global registry was limited to MACE (major adverse cardiac events) defined as the composite endpoint of death, myocardial infarction (Q- and non-Q-wave), emergent cardiac bypass surgery and TLR.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that results communications are provided to the sponsor at least 90 days prior to submittal for publication or presentation. The sponsor shall not require changes beyond the extent necessary to allow the sponsor to protect its rights in copyrightable material, and to check for technical correctness.